CLINICAL TRIAL: NCT01462331
Title: Double-blind, Randomized, Placebo Controlled Study to Investigate the Dietary Effects of VitaSugar/VitaFiber-IMO in Healthy Adults
Brief Title: the Dietary Effects of VitaSugar/VitaFiber-IMO in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioNeutra Inc. (Other)
Collaborators: Alberta Agriculture and Rural Development (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 11VBHB
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: Isomaltooligosaccharide; Human Consumption; Dose tolerance; Prebiotic; Short chain fatty acids; Blood glucose; Dose tolerance and prebiotic effect
MeSH Terms: interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- VitaSugar/VitaFiber-IMO dose-1 (Other): A group of 20 subjects (10 male and 10 females) will take IMO dose-1 (12g/dose) powder; three times a day dissolved in a glass of water
  Interventions: Other: Isomaltooligosaccharide (digestion-resistant carbohydrates)
- VitaSugar/VitaFiber-IMO dose-2 (Other): A group of 20 subjects (10 male and 10 females) will take IMO dose-2 (18g/dose) powder; three times a day dissolved in a glass of water
  Interventions: Other: Isomaltooligosaccharide (digestion-resistant carbohydrates)
- Placebo (Placebo Comparator): A group of 20 subjects (10 male and 10 females) will take Placebo (12g/dose) powder; three times a day dissolved in a glass of water
  Interventions: Other: Sucrose

INTERVENTIONS:
Other: Isomaltooligosaccharide (digestion-resistant carbohydrates) — 12g/dose; three times a day
  Other Names: VitaSugar; VitaFiber
  Arms: VitaSugar/VitaFiber-IMO dose-1
Other: Isomaltooligosaccharide (digestion-resistant carbohydrates) — 18g/dose, three times a day
  Other Names: VitaSugar; VitaFiber
  Arms: VitaSugar/VitaFiber-IMO dose-2
Other: Sucrose — 12g/dose, three times a day
  Other Names: Table top sugar
  Arms: Placebo

SUMMARY:
The purpose of this study is to re-confirm the already established health effects and dose tolerance of Isomalto-oligosaccharide or IMO, which is a general health/functional food ingredient.

DETAILED DESCRIPTION:
Isomalto-oligosaccharide (IMO) is a mixture of natural resistant carbohydrates consisting of short-chains of glucose molecules. IMO is made by enzymatic conversion of starch and uses as a health food ingredient with health benefits of a low calorie sweetener, prebiotic and dietary fiber. IMO have been ingested by humans for last many centuries as it is naturally found in rice miso, sake and soy sauce. IMO already got approval from FDA (GRAS) and from Health Canada.

There are number of published studies (in humans and animals) regarding the health benefits of IMO as an effective prebiotic, and its role in improving overall human gastric health. Studies also showed that IMO have found to be most tolerable with least adverse effects compared to other short-chain resistant oligosaccharides. Current clinical studies are conducted to verify the above given health benefits in BioNeutra's manufactured VitaSugar/VitaFiber-IMO products which including quantitative analysis of Bifidobacteria spp., Lactic acid bacteria group and clostridium spp. The production of short-chain fatty-acids (SCFA) and effect on blood glucose level are also analyzed in addition to the dose tolerance in term of lower and upper permissible dosage with resultant adverse effects if any are also observed.

ELIGIBILITY:
1. Male or female aged 18 to 65 years
2. If female, subject is not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation).

   OR

   Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:
   * Double-barrier method (condoms with spermicide or diaphragm with spermicide)
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Intrauterine devices
   * Vasectomy of partner
   * Abstinence
3. Healthy as determined by laboratory results, medical history
4. Agrees not to change current dietary habits and activity levels during the course of the study
5. Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
2. Participation in a clinical research trial within 30 days prior to randomization
3. History of or current diagnosis of any cancer (except for successfully treated basal cell carcinoma) diagnosed less than 5 years prior to screening. Subjects with cancer in full remission more than 5 years after diagnosis are acceptable.
4. Uncontrolled hypertension defined as untreated systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg or the use of medication for the treatment of hypertension
5. Unstable medications (dosage must be stable for 90 days prior to randomization
6. Clinically significant abnormal laboratory results at screening
7. History of gastrointestinal disease (appendectomy is acceptable) or diabetes
8. Use of antibiotics and/or laxatives within 2 months prior to randomization
9. Use of food or supplements containing probiotics within 2 weeks prior to randomization and during the course of the study
10. Alcohol or drug abuse in past year
11. Allergy or sensitivity to test product ingredients
12. Individuals who are cognitively impaired and/or who are unable to give informed consent
13. Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject Concomitant Medications Subjects will be required to washout for 14 days after taking any food or supplements containing probiotics before they can be randomized if the investigator determines that this will not negatively affect the subject's health. Subjects requiring prescribed medications for any acute or chronic conditions will be not be allowed to participate in this trial. Subjects cannot have used antibiotics or laxatives within the 2 months prior to randomization. Birth control is allowed during the study. Subjects who are currently taking prescribed birth control must agree to maintain their current method and dosing regimen during the course of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Dose Tolerance | one year
  To Evalaute the dietary effects of two dosages of VitaSugar/VitaFiber-IMO on digestive health in healthy adults.

SECONDARY OUTCOMES:
Effect of IMO on human colon microflora and clinical chemistry | One year
  To evaluate effect of VitaSugar/VitaFiber-IMO on human colon microflora and clinical chemistry, including: Prebiotic effect, Quantitative analysis of fecal samples for SCFA, Analysis of Glucose and insulin level and general clinical chemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Mal Evans, PhD, Principal Investigator — KGK Synergize
Locations (1):
- KGK Synergize, London, Ontario, Canada